CLINICAL TRIAL: NCT03457285
Title: A Feasibility Study to Investigate the Use of Salaso to Increase Access to Physiotherapy and Increase Compliance to Exercise Prescription and Physical Activity in the Management of Ankylosing Spondylitis (AS).
Brief Title: Investigating the Use of Salaso to Improve Physiotherapy Management of Ankylosing Spondylitis (AS).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. James's Hospital, Ireland (Other)
Collaborators: Salaso Health Solutions Limited (Unknown); Novartis (Industry)
Responsible Party: Principal Investigator, Ciaran Brennan, Senior Physiotherapist in Rheumatologuy, St. James's Hospital, Ireland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJH AS Salaso Study
Record Dates: First submitted 2018-02-01; First posted 2018-03-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing spondylitis; physiotherapy; Salaso
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: All participants will receive the same intervention
Masking Description: No masking will take place
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physiotherapy via the Salaso Apllication Intervention (Experimental): All participants' physiotherapy- prescribed exercise programmes will be monitored via the Salaso application. Telehealth appointments will occur monthly and modifications to exercises will be made as required.
  This will continue for the 6-month duration of the intervention.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Participants, with a confirmed diagnosis of AS, will be invited to participate. Once participants have provided informed consent, they will be required to complete the outcome measures provided. Participants will be set up to use the online exercise application and educated on its use.
  Participants will then have access to videos of suitable exercises or exercise classes to follow and education material on their condition to read. Participants will be able to complete AS specific outcome measures and record their progress. Participants will also have a monthly video call with the senior rheumatology physiotherapist to discuss their exercise programme, symptoms and management. The participants will also record their compliance with their exercise programmes.
  After the 6 month pilot period, participants will be required to complete the same outcome measures completed at the start of the study.
  Other Names: Salaso

SUMMARY:
This is a pilot study to investigate the use of Salaso, a web based exercise app, to increase access to physiotherapy and improve physical activity in patients attending St James's Hospital Rheumatology for Ankylosing Spondylitis (AS). Participants will be set up on the app and given an individual exercise programme. All individual exercises and exercise class videos will be available on the app. Completion of exercises can be logged on the app and exercise compliance will then be monitored remotely by the physiotherapist through the Salaso app. The physiotherapist will have a monthly telehealth session with each participant to assess progress and to address any difficulties. Outcome measures will be completed at initial assessment and again at the end of the pilot study. This data will then be analysed to assess the effectiveness of the Salaso app as a treatment option for AS.

DETAILED DESCRIPTION:
AS is a chronic inflammatory condition affecting the spine and other joints, causing pain and stiffness. Currently approximately 150 people attend Saint James's Hospital rheumatology department for management of their condition. Physiotherapy plays a key role in this management. As this is often a younger patient population, it can be challenging for them to attend appointments due to work and family commitments. It is envisaged that this pilot will enhance treatment options for all participants.

The aims of this study are: to improve use of exercise and physical activity using an online exercise application; to improve self-management skills in monitoring progress and ability to exercise independently using an online exercise application; to provide an online appointment review option to patients who are unable to attend physiotherapy appointments in St James's Hospital.

Descriptive statistics will be used to record and analyse the study data, using SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Ankylosing Spondylitis

Exclusion Criteria:

* Previous spinal surgery
* Spondylolisthesis
* Unwillingness to participate
* Unable to complete self-report questionnaires
* Progressive neurological deficit
* Neurological disease
* Cauda equina syndrome
* Unable to exercise on medical grounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-17 (Actual); Primary Completion 2019-04-17 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Bath Ankylosing Spondylitis Metrology Index | 6 months
  Measure of spinal mobility

SECONDARY OUTCOMES:
Bath Ankylosing Spondylitis Disease Activity Index | 6 months
  Measuring disease activity in AS
Bath Ankylosing Spondylitis Functional Index | 6 months
  Measuring functional activity in AS
Arthritis Self-Efficacy Scale (ASES) | 6 months
  The scale is an assessment of a person's ability to self-manage his/her pain, function and other symptoms. The self-efficacy function scale has 9 questions, each scored on a scale of 1-10, with a total minimum score of 10 and a maximum score of 90. The self-efficacy pain scale has 5 questions, with a total minimum score of 5 and a maximum score of 50. The self-efficacy other symptoms scale has 6 questions, with a minimum total score of 6 and a maximum score of 60. The other symptoms scale and the pain scale may be combined, with a sum score given.
Exercise Benefits/Barriers Scale (EBBS) | 6 months
  Measuring the perceived benefits of and barriers to performing the prescribed exercises. There are 43 questions in total. It may be scored in it's entirety or as two separate scales. Scores can range from 43 to 172. The higher the score, the more positively the individual perceives exercise. The benefits scale is scored between 29 and 116. The barriers scale is scored between 14 and 56. The higher the score on the barriers scale, the greater the perception of barriers to exercise. If combined, the barriers scale is reverse-scored.

CONTACTS AND LOCATIONS:
Overall Officials: Finbar O'Shea, Principal Investigator — Consultant Rheumatologist, Saint James's Hospital
Locations (1):
- Physiotherapy Department, Saint James's Hospital, Dublin, Ireland